CLINICAL TRIAL: NCT00847483
Title: A Comparison of Latanoprost (Xalatan) With Travoprost (Travatan) and Bimatoprost (Lumigan) in Patients With Elevated Intraocular Pressure. A Twelve-week, Masked Evaluator, Phase IV, Multicenter Study in the United States. (Xalatan vs Travatan vs Lumigan).
Brief Title: Comparison of Latanoprost With Travoprost and Bimatoprost in Patients With Elevated IOP. A 12-weeks, Masked Evaluator, Phase IV Multi-center Study in the US
Acronym: XLT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XALA-0091-157; A6111081
Record Dates: First submitted 2009-02-16; First posted 2009-02-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2009-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular hypertension; latanoprost; travoprost; bimatoprost
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; Ophthalmic Solutions; Travoprost; Bimatoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Latanoprost (Active Comparator)
  Interventions: Drug: latanoprost 0.005% ophthalmic solution
- Travoprost (Active Comparator)
  Interventions: Drug: Travoprost 004% sterile ophthalmic solution
- Bimatoprost (Active Comparator)
  Interventions: Drug: Bimatoprost .03% sterile ophthalmic solution

INTERVENTIONS:
Drug: latanoprost 0.005% ophthalmic solution — One drop in the evening in the affected eye(s) at 8:00pm
  Other Names: Xalatan
  Arms: Latanoprost
Drug: Travoprost 004% sterile ophthalmic solution — One drop in the evening in the affected eye(s) at 8:00pm
  Other Names: Travatan
  Arms: Travoprost
Drug: Bimatoprost .03% sterile ophthalmic solution — One drop in the evening in the affected eye(s) at 8:00pm
  Other Names: Lumigan
  Arms: Bimatoprost

SUMMARY:
Compare the IOP lowering properties of latanoprost, travoprost and bimatoprost

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary open angle glaucoma (POAG), exfoliative glaucoma, pigmentary glaucoma or ocular hypertension (glaucoma is defined as either visual fields defect or glaucomatous changes of the optic nerve head in association with elevated intraocular pressure. Ocular hypertension is defined as IOP ≥ 21 mmHg at diagnosis).
* Is currently receiving (at the screen visit) or has received topical monotherapy or dual therapy (within the past 6 months) for POAG or ocular hypertension.
* Required washout periods are 4 weeks for -adrenergic antagonists, prostaglandin analogues (including latanoprost, unoprostone, travoprost and bimatoprost) and 2 weeks for adrenergic agonists, and 5 days for cholinergic agonists and carbonic anhydrase inhibitors, prior to the baseline visit.
* Mean 8 AM IOP ≥ 23 mmHg at the baseline visit for all patients. Patients should be assigned treatment only after the 8 PM IOP is obtained.
* Visual acuity (best corrected) equal to or better than 20/200 (Snellen). ETDRS charts may be used and converted to Snellen units.
* Informed Consent: Signed Informed Consent is obtained at the screen visit.
* Able to adhere to treatment/visit planUnilateral or bilateral primary open angle glaucoma, capsular glaucoma, pigmentary glaucoma or ocular hypertension.
* Open angle glaucoma appearing more than 6 months after cataract surgery is recognized as primary open angle glaucoma. (individuals requiring treatment bilaterally must fulfill eligibility criteria for both eyes.)
* IOP of 22mmHg or higher obtained during the pre-study period.

Exclusion Criteria:

Ocular conditions

* Closed/barely open anterior chamber angle or history of acute angle closure. (Patients who are diagnosed with POAG after a successful peripheral iridotomy may be enrolled).
* History of ALT (Argon Laser Trabeculoplasty) within 3 months prior to the screen visit (the unlasered eye may be enrolled as the study eye).
* History of any ocular filtering surgical intervention (the unfiltered eye may be enrolled as the study eye).
* Ocular surgery (on the globe of the eye only), or inflammation/infection within 3 months prior to screen visit. (Applies to both fellow and study eyes.)
* Hypersensitivity to benzalkonium chloride or to any other component in latanoprost (Xalatan), travoprost (Travatan) or bimatoprost (Lumigan).
* Other abnormal ocular conditions or symptoms preventing the patient from entering the study, in the investigator's clinical judgement.

Other conditions

* Use of systemic medication known to affect IOP (i.e., alpha-adrenergic agonists, beta-adrenergic antagonists, calcium channel blockers, ACE inhibitors and/or angiotensin II receptor blockers, or corticosteroids), unless the patient and the medication dosage have been stable for three months prior to the screen visit and the dosage is not expected to change during the study.

Women

* Women of childbearing potential (WOCBP) who are not using contraceptive methods. Women of childbearing potential are defined as women who are not surgically sterile or not postmenopausal (at least 12 months without a menstrual period). Contraception is defined as abstinence, having a vasectomized partner, or the ongoing use of approved oral, injectable or implanted contraceptives, a barrier method, or an IUD.
* Pregnancy. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at the screen visit and baseline visit.
* Nursing mothers General
* Use of any investigational medication within 30 days prior to screen visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2002-01; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
To compare the IOP reducing effect of latanoprost (Xalatan) versus travoprost (Travatan) versus bimatoprost (Lumigan) over a twelve-week period. | 12 weeks
The mean change since baseline of Week 12 IOP measured at the time of peak (8:00AM) drug effect. | 12 weeks

SECONDARY OUTCOMES:
To study the safety variables within and between all treatment groups over 12 weeks | 12 weeks
The mean change since baseline of Week 12 IOP measured at the time of trough (8:00PM) drug effect. The mean percentage change since baseline of diurnal IOP at Week 12. | 12 weeks
The mean change since baseline of Week 12 IOP measured at the times of peak (8:00AM) and trough (8:00PM) drug effects evaluated by race. The percentage of patient withdrawals from the study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (34):
  - Pfizer Investigational Site, Bellflower, California
  - Pfizer Investigational Site, Inglewood, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Bloomingdale, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Bangor, Maine
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Bloomfield, New Jersey
  - Pfizer Investigational Site, Willingboro, New Jersey
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Streetsboro, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Maryville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Wenatchee, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XALA-0091-157&StudyName=Comparison%20of%20latanoprost%20with%20travoprost%20and%20bimatoprost%20in%20patients%20with%20elevated%20IOP.%20A%2012-weeks%2C%20masked%20evaluator%2C%20phase%20IV%20m